CLINICAL TRIAL: NCT04292756
Title: Safety and Effectiveness of Triamcinolone Acetonide in Patients With Serous Pigment Detachment Associated With Age-Related Macular Degeneration
Brief Title: Triamcinolone Acetonide in Patients With Serous Pigment Epithelial Detachment
Acronym: COAST_UA_AMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Filatov Institute of Eye Diseases and Tissue Therapy (Other)
Collaborators: Odessa National Medical University (Other); Mykolaiv Region Ophthalmogical Hospital (Other); Central Polyclinic of Internal Affairs of Ukraine (Other Government)
Responsible Party: Principal Investigator, Andrii Korol, MD, PhD, Head of Laser Department, The Filatov Institute of Eye Diseases and Tissue Therapy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0118U001612/4
Record Dates: First submitted 2020-02-28; First posted 2020-03-03 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Age-Related Macular Degeneration
Keywords: Age-related macular degeneration; serous pigment epithelium detachment; triamcinolone acetonide
MeSH Terms: conditions — Macular Degeneration | interventions — Triamcinolone Acetonide; Fluorescein Angiography; Slit Lamp Microscopy; Ophthalmoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Triamcinolone Acetonide 40 mg (Active Comparator): Arm 1
  Interventions: Procedure: Subtenon injection of 40 mg triamcinolone acetonide; Diagnostic Test: Visometry; Diagnostic Test: Fluorescent angiography; Diagnostic Test: Refractometry; Diagnostic Test: Slit lamp examination; Diagnostic Test: Ophthalmoscopy; Diagnostic Test: OKT; Diagnostic Test: IOP
- Triamcinolone Acetonide 4 mg (Active Comparator): Arm 2
  Interventions: Procedure: Intravitreal injection of 4 mg triamcinolone acetonide; Diagnostic Test: Visometry; Diagnostic Test: Fluorescent angiography; Diagnostic Test: Refractometry; Diagnostic Test: Slit lamp examination; Diagnostic Test: Ophthalmoscopy; Diagnostic Test: OKT; Diagnostic Test: IOP

INTERVENTIONS:
Procedure: Subtenon injection of 40 mg triamcinolone acetonide — Subtenon injection of 40 mg triamcinolone acetonide: 1 initial injection of 40 mg triamcinolone acetonide, further injections will be base at month 3 examination.
  Arms: Triamcinolone Acetonide 40 mg
Procedure: Intravitreal injection of 4 mg triamcinolone acetonide — Intravitreal injection of 4 mg triamcinolone acetonide: 1 initial injection of 4 mg triamcinolone acetonide, further injections will be base at month 3 examination.
  Arms: Triamcinolone Acetonide 4 mg
Diagnostic Test: Visometry — Ophthalmic examination
Diagnostic Test: Fluorescent angiography — Ophthalmic examination
Diagnostic Test: Refractometry — Ophthalmic examination
Diagnostic Test: Slit lamp examination — Ophthalmic examination
Diagnostic Test: Ophthalmoscopy — Ophthalmic examination
Diagnostic Test: OKT — Ophthalmic examination
Diagnostic Test: IOP — Ophthalmic examination

SUMMARY:
The purpose of this study is to determine the effectiveness and safety of triamcinolone acetonide in patients with serous pigment detachment associated with age-related macular degeneration

DETAILED DESCRIPTION:
The purpose of this study is to determine the effectiveness and safety of triamcinolone acetonide in patients with serous pigment epithelial detachment associated with age-related macular degeneration.

This study is planned as a follow-up. Patients with with serous pigment epithelial detachment associated with age-related macular degeneration included in it will receive triamcinolone acetonide in accordance with the approved indications for use indicated in the instructions for the use of drugs in Ukraine.

The treatment proposed in this study is based on the world experience and scientific developments of the Filatov Institute of Eye Diseases and Tissue Therapy of the NAMS of Ukraine ". Therefore, it is expected that the benefit / risk ratio in relation to the participation in this study should not be different from that described in the scientific literature and the benefits outweigh the risk. It is known that the absence of treatment in these diseases leads to an irreparable loss of central vision.

ELIGIBILITY:
Inclusion Criteria:

* Able to read (or, if unable to read due to visual impairment, be read to verbatim by the person administering the informed consent form or a family member) and understand the informed consent form and willing to sign the informed consent form.
* Signed informed consent form.
* Men and women ≥ 50 years of age.
* Willing, committed, and able to return for all clinic visits and complete all study-related procedures.
* Naive serous pigment epithelial detachment associated with AMD as defined on FA and OCT.
* Transparent optical media and possibility to mydriasis.
* Best corrected visual acuity at least 20/100 Equivalent of Snellen (ETDRS).
* Absence of signs of CNV, angiomatous retina proliferation, polypoid choriovasculopathy defined on FA and OCT.

Exclusion Criteria:

* Ocular media of insufficient quality to obtain fundus and OCT images in the study eye.
* Previous intravitreal injections of anti-VEGF drugs in the study eye.
* Any injections of corticosteroids (intravitreal, subtenon, subconjunctival or parabulbar) or implantation of medical device in the study eye.
* Ocular inflammation or external ocular inflammation in the study eye.
* Concurrent disease in the study eye that would compromise BCVA or require medical or surgical intervention during the study period.
* Any ocular disorder in the study eye that, in the opinion of the investigator, may confound interpretation of the study results.
* Significant scarring or atrophy in the fovea that indicates substantial irreversible vision loss in the study eye.
* Evidence at examination of infectious blepharitis, keratitis, scleritis, or conjunctivitis in either eye or current treatment for serious systemic infection.
* Vitreomacular traction or traction retinal detachment, epiretinal membrane in study eye.
* Any iris neovascularization and/or vitreous hemorrhage in either eye.
* Uncontrolled glaucoma, or previous filtration surgery in either eye.
* Maсular hole.
* Any prior treatment with photodynamic therapy in the study eye.
* Cataract surgery within 3 months prior to Day 1 in the study eye.
* Yttrium-aluminum-garnet laser capsulotomy within 2 months prior to Day 1 in the study eye.
* Any other intraocular surgery within 3 months prior to Day 1 in the study eye.
* History of vitreoretinal surgery and/or scleral buckle surgery in the study eye.
* Previous assignment to treatment during this study.
* Uncontrolled hypertension.
* History of cerebrovascular disease or myocardial infarction within 6 months prior to Baseline/Day 1.
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug, may affect interpretation of the results of the study, or renders the subject at high risk from treatment complications.
* Women of childbearing potential without contraception, women who intend to breastfeed during the study. All subjects (both men and women) of childbearing potential who are unwilling to use adequate birth control measures during the course of the study.
* Renal failure requiring dialysis or renal transplant.
* Participation in an investigational study within 30 days prior to Screening/Visit 1 that involved treatment with any drug (excluding vitamins and minerals) or device.
* Known serious allergy to the fluorescein sodium for injection in angiography or Verteporfin.
* Inability to obtain fundus photographs or fluorescein angiograms of sufficient quality.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Mean Change in Best Corrected Visual Acuity (BCVA) as Measured by ETDRS Chart | Baseline-Month 12
  Defined study baseline range of ETDRS equivalent of 20/200 to 20/20) in the study eye; a higher score represents better functioning.

SECONDARY OUTCOMES:
Number of Flattened Pigment Epithelial Detachment | Baseline-Month 12
  Number of flattened pigment epithelial detachment
Mean Change in Central Retinal Thickness (CRT) as Assessed by Optical Coherence | Baseline-Month 12
  A negative number indicates improvement (reduced thickness).
Average Number of Injections | Baseline-Month 12
  The number of injections administered
Intraocular pressure | Baseline-Month 12
  The difference between intraocular pressure at baseline and at Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Andrii MD Korol, PhD, Principal Investigator — The Filatov Institute of Eye Diseases and Tissue Therapy
Locations (4):
- Ukraine (4):
  - Odessa National Medical University, Odesa, Please Select
  - CPUkraine, Kyiv
  - Mykolaiv Region Ophthalmogical Hospital, Mykolaiv
  - The Filatov Institute of Eye Diseases and Tissue Therapy, Odesa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] V Pasyechnikova N, A Naumenko V, R Korol A, S Zadorozhnyy O, B Kustrin T, O Nasinnyk I. Serous pigment epithelium detachment associated with age-related macular degeneration: a possible treatment approach. Med Hypothesis Discov Innov Ophthalmol. 2012 Winter;1(4):72-5. PMID 24600628